CLINICAL TRIAL: NCT02045160
Title: A Pharmacokinetic and Pharmacogenetic Study in Patients Receiving Sulfamethoxazole-trimethoprim Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 201312090RINC
Record Dates: First submitted 2014-01-17; First posted 2014-01-24 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Pneumocystis Jirovecii Pneumonia
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Sulfamethoxazole-trimethoprim treatment

SUMMARY:
In this study, we aim to investigate the incidence of the adverse reactions, the effectiveness and the gene polymorphism associated with the plasma level of sulfamethoxazole-trimethoprim and their metabolites (including N4-acetyl-sulfamethoxazole, sulfamethoxazole hydroxylamine and sulfamethoxazole-nitroso). And we also aim to investigate the factors associated with the sulfamethoxazole-trimethoprim induced acute psychosis.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 20 years or older
* using oral or intravenous form of sulfamethoxazole-trimethoprim

Exclusion Criteria:

* patients who are under 20 years of age

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated in the National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
High performance liquid chromatography for drug plasma concentration | Participants will be followed for the duration of the treatment course, an expected average of 21 days
  The plasma concentration will not be measured until the patient's treatment course completed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, TW, Taiwan